CLINICAL TRIAL: NCT06504966
Title: A Randomized, Double-blind, Parallel-group, Active-controlled Study to Compare the Efficacy, Pharmacokinetics, Pharmacodynamics, Safety, and Immunogenicity of MAB-22 Versus Prolia® Sourced From the European Union in Postmenopausal Women With Osteoporosis
Brief Title: Study to Compare the Efficacy, Pharmacokinetics, Pharmacodynamics, Safety, and Immunogenicity of MAB-22 Versus Prolia®
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Business decision not to proceed with the study.
Sponsor: Xentria, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: MAB-22-301
Record Dates: First submitted 2024-07-10; First posted 2024-07-17 (Actual); Last update posted 2025-05-11 (Actual); Status verified 2024-11

CONDITIONS: Osteoporosis
MeSH Terms: conditions — Osteoporosis | interventions — Denosumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Double Blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- MAB-22 (Experimental): Single subcutaneous dose at Day 1 (baseline), 6 months (Week 26) and Visit 12 (Week 52)
  Interventions: Drug: MAB-22
- Prolia® and MAB-22 (Experimental): Single subcutaneous dose of Prolia® at Day 1 (baseline), 6 months (Week 26) and single subcutaneous dose of MAB-22 (switching) or Prolia ® (non-switching) at Visit 12 (Week 52)
  Interventions: Drug: MAB-22; Drug: Prolia®

INTERVENTIONS:
Drug: MAB-22 — Single subcutaneous dose of 60 mg
Drug: Prolia® — Single subcutaneous dose of 60 mg
  Arms: Prolia® and MAB-22

SUMMARY:
Double-blind, Parallel-group, Active-controlled Study to Compare the Efficacy, Pharmacokinetics, Pharmacodynamics, Safety, and Immunogenicity of MAB-22 Versus Prolia®

DETAILED DESCRIPTION:
A Randomized, Double-blind, Parallel-group, Active-controlled Study to Compare the Efficacy, Pharmacokinetics, Pharmacodynamics, Safety, and Immunogenicity of MAB-22 Versus Prolia® Sourced from the European Union in Postmenopausal Women with Osteoporosis

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent must be obtained before participation in the study.
2. Postmenopausal women diagnosed with osteoporosis (consistent with a lumbar spine bone mineral density (LS-BMD) [L1-L4] or TH-BMD T-score of ≤ -2.5 and ≥ -4.0 as measured by dual x-ray absorptiometry (DXA) at screening). Postmenopausal status is defined as at least 12 consecutive months of amenorrhea before date of screening, for which there is no other obvious pathological or physiological cause.
3. Between ≥55 and ≤80 years of age at screening.
4. Body weight ≥50 kg and ≤90 kg at screening.
5. At least 3 vertebrae in the L1-L4 region (vertebrae to be assessed by local reading of lateral spine x-ray at screening) and at least one hip joint are evaluable by DXA.
6. Adequate organ function as defined by the following criteria:

   1. Serum aspartate aminotransferase (AST) and serum alanine aminotransferase (ALT) ≤2.5 × upper limit of normal (ULN).
   2. Total serum bilirubin ≤1.5 × ULN.
   3. Absolute neutrophil count ≥1500 cells/μL (SI units: ≥1.5 × 109/L).
   4. Platelet count ≥100,000 cells/μL (SI units: ≥100 × 109/L) and ≤ULN.
   5. Hemoglobin ≥10 g/dL and ≤ULN.
   6. Albumin-adjusted serum calcium within the normal range for the testing laboratory.
   7. Estimated glomerular filtration rate >45 mL/min.

Exclusion Criteria:

1. Previous exposure to denosumab (Prolia®, Xgeva®, or biosimilar denosumab).
2. History of hypersensitivity to any recombinant protein drugs or any of the excipients used in MAB-22 or Prolia®.
3. History and/or presence of 1 severe or more than 2 moderate vertebral fractures or hip fractures (as determined by local reading of lateral spine x-ray at screening). Osteoporotic-related fracture (i.e., crush or wedge vertebral fracture or hip fracture) known or suspected to have occurred within 6 months of randomization.
4. Recent long bone fracture (within 6 months) before screening. Presence of active healing fracture according to assessment of investigators.
5. History and/or presence of bone metastases, bone disease, or metabolic disease, other than osteoporosis, which could interfere with the interpretation of the findings (e.g., osteogenesis imperfecta, osteopetrosis, osteomalacia, rheumatoid arthritis, Paget's disease, ankylosing spondylitis, Cushing's disease, hyperprolactinemia, malabsorption syndrome, hypoparathyroidism or hyperparathyroidism [irrespective of current controlled or uncontrolled status], hypocalcemia or hypercalcemia [based on albumin-adjusted serum calcium]).
6. Malignancy within the 5 years before screening (except cervical carcinoma in situ or basal cell carcinoma, which are acceptable).
7. Ongoing use of any osteoporosis treatment (other than calcium and vitamin D supplements). The following rules for washout periods for osteoporosis treatments must be adhered to:

   1. Drugs being investigated for osteoporosis (e.g., romosozumab): dose received at any time.
   2. Strontium or fluoride (for osteoporosis): dose received at any time.
   3. Tibolone, oral or transdermal estrogen, selective estrogen receptor modulators, systemic hormone replacement therapy: dose received within 12 months before screening.
   4. Calcitonin, calcitriol, maxacalcitol, falecalcitriol, or alfacalcidol: dose received within 3 months before screening.
   5. Cinacalcet: dose received within 3 months before screening.
   6. Any oral bisphosphonate treatment. Note: those participants who have taken oral bisphosphonates for up to 3 months, or >3 months but <3 years cumulatively are eligible after a 12-month washout period.
   7. Intravenous bisphosphonates: dose received within 5 years before the first administration of study treatment.
   8. Parathyroid hormone (PTH), or PTH derivatives within the last 12 months before the first administration of study treatment.
8. Other bone active drugs including heparin, anti-convulsives (with the exception of benzodiazepines), systemic ketoconazole, adrenocorticotropic hormone, lithium, gonadotropin releasing hormone agonists, and anabolic steroids, within the past 3 months before the first administration of study treatment.
9. Systemic glucocorticosteroids (≥5 mg prednisone equivalent per day for ≥10 days or a total cumulative dose of ≥50 mg) within the past 3 months before screening.
10. Use of other investigational drugs within 2 months of screening (or 5 half-lives of the drug or until the expected Pharmacodynamic (PD) effect of the drug has returned to baseline, whichever is longer) or longer if required by local regulations.
11. Oral or dental conditions: osteomyelitis or history and/or presence of osteonecrosis of the jaw (ONJ), presence of risk factors for ONJ (e.g., periodontal disease, poorly fitting dentures, invasive dental procedures such as tooth extractions in 6 months before screening), active dental or jaw condition which requires oral surgery and/or planned invasive dental procedure.
12. Recent tooth extraction (within 6 months of the screening visit). Edentulous participants are permitted to enroll in the study, as long as the most recent tooth extraction occurred >6 months of the screening visit.
13. Vitamin D deficiency (25-[OH] vitamin D serum level <20 ng/mL). Vitamin D repletion is permitted at the discretion of the investigator, and participants will be rescreened to reevaluate vitamin D level post-repletion.
14. Known intolerance to, or malabsorption of calcium or vitamin D supplements.
15. History and/or presence of a severe allergic reaction (e.g., anaphylaxis).
16. Has a hepatitis B surface antigen, hepatitis C antibody, or human immunodeficiency virus (HIV) antibody positive at screening.
17. History and/or presence of significant cardiac disease as per investigator's discretion, including but not restricted to: Electrocardiogram (ECG) abnormalities at screening indicating significant risk of safety for participants participating in the study, history and/or presence of myocardial infarction within 6 months before screening, history and/or presence of New York Heart Association (NYHA) class III or IV heart failure.
18. History of prior allogeneic transplantation.
19. Have a history of alcohol or drug abuse in the judgment of the investigator within the previous 12 months before screening.
20. Unstable systemic disease including active infection, uncontrolled hypertension, unstable angina, congestive heart failure, or myocardial infarction within 6 months before randomization.
21. Have major surgery (including surgery to bone), or significant traumatic injury occurring within 4 weeks before randomization.

Ages: 55 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-10 (Estimated); Primary Completion 2027-10 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
To compare MAB-22 and Prolia® (EU-authorized) in postmenopausal women with osteoporosis to demonstrate biosimilarity and non-inferiority with respect to efficacy profile in terms of bone mineral density (BMD). | Day 1 to Week 52
  Efficacy coprimary endpoint: percentage change from baseline (%CfB) in lumbar spine bone mineral density (BMD) (LS-BMD)
To compare MAB-22 and Prolia® (EU-authorized) in postmenopausal women with osteoporosis to demonstrate biosimilarity and non-inferiority with respect to Pharmacodynamic (PD) profile in terms of serum cross-linked C telopeptide of type I collagen (sCTX). | Day 1 to Week 26 [Predose]
  PD coprimary endpoint: area under the effect curve (AUEC) of C telopeptide of type I collagen (sCTX) over the initial 6-month period

IPD SHARING:
Plan to Share IPD: No